CLINICAL TRIAL: NCT02741908
Title: Effects of Two Diet Techniques and Delivery Mode on Weight Loss, Metabolic Profile and Food Intake of Obese Adolescents: a Fixed Diet Plan and a Calorie Counting Diet
Brief Title: Fixed Diet Plan and Calorie Counting Diet in Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MARCIO CORRÊA MANCINI (Other)
Responsible Party: Sponsor-Investigator, MARCIO CORRÊA MANCINI, Head of the Obesity and Metabolic Syndrome Unit at the Department of Endocrinology and Metabolism, University of Sao Paulo
Organization: University of Sao Paulo (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0037/11
Record Dates: First submitted 2016-04-13; First posted 2016-04-18 (Estimated); Last update posted 2016-04-18 (Estimated); Status verified 2016-04

CONDITIONS: Pediatric Obesity
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fixed diet plan (Experimental): Patients received a fixed diet plan to assist in the choice of foods aimed at changing eating behavior. Dietary intake was evaluated by using 3 nonconsecutive 24-hour dietary recalls collected at each visit. Received a reduction of 500 calories in the total energy expenditure calculated by the equation predicted by Dietary Reference Intake (DRI) from the Institute of Medicine (2005). Also received qualitative information regarding healthy food behaviours, by a same dietitian, based on the DRI for Acceptable Macronutrient Ranges, appropriated for age and gender.
  Interventions: Behavioral: Fixed diet plan
- Calorie counting diet (Experimental): Patients underwent a calorie counting diet, in which each patient has received a table list with equivalent points for food and drinks, and was instructed to record all daily food or drink intake and calculate the total score of points consumed (1 point = 3.6 calories). They were allowed to eat any food but were limited to the recommended amount of points (or calories equivalents). Received a reduction of 500 calories in the total energy expenditure calculated by the equation predicted by Dietary Reference Intake (DRI) from the Institute of Medicine (2005). Also received qualitative information regarding healthy food behaviours, by a same dietitian, based on the DRI for Acceptable Macronutrient Ranges, appropriated for age and gender.
  Interventions: Behavioral: Calorie counting diet

INTERVENTIONS:
Behavioral: Calorie counting diet
  Arms: Calorie counting diet
Behavioral: Fixed diet plan
  Arms: Fixed diet plan

SUMMARY:
Obesity is a chronic illness and multifactorial etiology, related to genetic factors, environmental and behavioral. Features association with several metabolic abnormalities in childhood, leading to increased risk of cardiovascular disease in adult life. The treatment involves lifestyle change, with balanced diet guidance and encouraging physical activity. The treatment in this age group have brought limited data, in addition to high drop-out rates. A unique type of food guidance is the equivalent calorie count, where calories are converted into points. The objective of this study was to evaluate the variance of Z score of body mass index (ZIMC) of obese adolescents undergoing orientation of two groups of low-calorie diet: traditional and based on the points system, as well as evaluate anthropometric variables, body composition, food intake, metabolic changes and self-monitoring.

METHODS: randomized clinical study with duration of 24 weeks, with 66 adolescents with an average age of 13.7 ± 0.7 years of both genders, with scores of BMI >= 2 to <= 4 curve adjusted for gender and age of the World Health Organization. Were verified weight, height, blood pressure and waist circumference, intensity of physical activity and self- monitoring, as well as performed the nutritional guidance to each visit. Laboratory parameters, applying the scale of binge eating, pubertal, stage and body composition were evaluated at the beginning and end of the action. The patients were divided into two groups: one that received guidance of traditional low-calorie diet and meet the food consumption record (RCA), three days (Group A) and another that received low-calorie diet guidance based on the system of points and meet the daily RCA (Group B).

ELIGIBILITY:
Inclusion Criteria:

* Age 12 to 15 years old
* ZBMI ≥+2.0 according to World Health Organization

Exclusion Criteria:

* ZBMI≥+4
* obesity related to genetic syndromes
* End-organ damage
* Taking drugs that promote weight changes

Ages: 12 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 66 (Actual)
Dates: Start 2011-07; Primary Completion 2013-06 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Z-score body mass index | 24 weeks

IPD SHARING:
Plan to Share IPD: No